CLINICAL TRIAL: NCT00969436
Title: A Phase IIIb, Open, Randomised, Multicentre, Primary Study in Healthy Children, to Establish the Non-inferiority of GlaxoSmithKline (GSK) Biologicals' MeMuRu-OKA Vaccine (Administered at 9 and 15 Months of Age) Versus Priorix™ (9 Months of Age) and Priorix™ Co-administered With Varilrix™ at 15 Months of Age (Comparator) and Also to Evaluate the Non-inferiority of Priorix™ (9 Months of Age) and MeMuRu-OKA Vaccine (15 Months of Age) Versus the Comparator, All Administered Subcutaneously as Two-dose Primary Vaccination Course
Brief Title: Comparison of GSK Measles-mumps-rubella-varicella (MMRV) Vaccine Versus PriorixTM
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 109995
Record Dates: First submitted 2009-08-20; First posted 2009-09-01 (Estimated); Results first posted 2017-09-25 (Actual); Last update posted 2018-06-08 (Actual); Status verified 2017-05

CONDITIONS: Varicella; Rubella; Mumps; Measles
Keywords: Mumps; Immunogenicity; Vaccines; Safety; Rubella; Combined Vaccine; Varicella Vaccine; Children; Measles; Humans
MeSH Terms: conditions — Chickenpox; Rubella; Mumps; Measles | interventions — Measles-Mumps-Rubella Vaccine

ARMS (3):
- Priorix-Tetra Group (Experimental): Subjects received 2 doses of Priorix-Tetra® vaccine, 1 at Day 0 and 1 at Month 6, administered subcutaneously in the left anterolateral thigh.
  Interventions: Biological: GSK Biological's investigational MMRV vaccine 208136
- Priorix/ Priorix-Tetra Group (Experimental): Subjects received 1 dose of Priorix™ vaccine at Day 0 and 1 dose of Priorix-Tetra® vaccine at Month 6, both administered subcutaneously in the left anterolateral thigh.
  Interventions: Biological: GSK Biological's investigational MMRV vaccine 208136; Biological: Priorix™
- Control Group (Active Comparator): Subjects received 1 dose of Priorix™ vaccine at Day 0 and 1 dose of Priorix™ vaccine co-administered with Varilirix™ vaccine at Month 6, administered subcutaneously in the left and right anterolateral thigh.
  Interventions: Biological: Priorix™; Biological: Varilrix™

INTERVENTIONS:
Biological: GSK Biological's investigational MMRV vaccine 208136 — Subcutaneous injection
  Arms: Priorix-Tetra Group; Priorix/ Priorix-Tetra Group
Biological: Priorix™ — Subcutaneous injection
  Arms: Control Group; Priorix/ Priorix-Tetra Group
Biological: Varilrix™ — Subcutaneous injection
  Arms: Control Group

SUMMARY:
The purpose of this study is to assess non-inferiority of two different vaccination regimens using GSK Biological's MMRV vaccine (two doses at 9 and 15 months) or Priorix™ (9 months) and one dose of MMRV vaccine (15 months) to the current standard of care which is Priorix™ administered at 9 months of age followed by concomitant administration of Priorix™ with Varilrix™ at 15 months of age in a measles endemic environment such as India.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes that their parents/guardians can and will comply with the requirements of the protocol should be enrolled in the study.
* Male or female subjects between and including 9 and 10 months of age at the time of the first vaccination.
* Written informed consent obtained from the the parent or guardian of the subject.
* Healthy subjects as established by medical history and clinical examination before entering into the study.

Exclusion Criteria:

* Use of any investigational or non-registered product other than the study vaccines within 30 days preceding the first dose of study vaccine, or planned use during the study period.
* Chronic administration of immunosuppressants or other immune-modifying drugs within six months prior to the first vaccine dose.
* Planned administration/administration of a vaccine not foreseen by the study protocol starting 30 days prior to administration of any dose of the study vaccine, up to 42 days after the vaccine dose with the exception of hepatitis A vaccine and oral poliovirus vaccine .
* Concurrently participating in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-registered product.
* Previous vaccination against measles, mumps, rubella and varicella.
* History of measles, mumps, rubella and/or varicella diseases.
* Known exposure to measles, mumps, rubella and/or varicella within 30 days prior to the start of the study.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination.
* A family history of congenital or hereditary immunodeficiency.
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccines including neomycin.
* Major congenital defects or serious chronic illness.
* History of any neurologic disorders or seizures.
* Acute disease at the time of enrolment.
* Axillary temperature > 37.5°C (99.5°F) / Rectal temperature > 38°C (100.4°F).
* Administration of immunoglobulins and/or any blood products during the six months before entering the study or planned administration during the study period.
* Presence of a susceptible high-risk person in the same household during the study period.

Ages: 9 Months to 10 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 450 (Actual)
Dates: Start 2009-11-09 (Actual); Primary Completion 2011-02-21 (Actual); Study Completion 2011-02-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (5):
- India (5):
  - GSK Investigational Site, Bangalore
  - GSK Investigational Site, Chennai
  - GSK Investigational Site, Goa
  - GSK Investigational Site, Kolkata
  - GSK Investigational Site, Pune

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Lalwani S, Chatterjee S, Balasubramanian S, Bavdekar A, Mehta S, Datta S, Povey M, Henry O. Immunogenicity and safety of early vaccination with two doses of a combined measles-mumps-rubella-varicella vaccine in healthy Indian children from 9 months of age: a phase III, randomised, non-inferiority trial. BMJ Open. 2015 Sep 11;5(9):e007202. doi: 10.1136/bmjopen-2014-007202. PMID 26362659
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Study Protocol: 109995 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 109995 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 109995 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 109995 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 109995 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 109995 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 109995 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: During the screening the following steps occurred: check for inclusion/exclusion criteria, contraindications/precautions, medical history of the subjects and signing informed consent forms.
Period: Overall Study
Arm/Group | Priorix-Tetra Group | Priorix/ Priorix-Tetra Group | Control Group
Started | 180 | 180 | 90
Completed | 155 | 159 | 79
Not Completed | 25 | 21 | 11
Not completed — Protocol Violation | 1 | 3 | 0
Not completed — Migrated/moved from study area | 12 | 10 | 2
Not completed — Father - serious health problem | 0 | 0 | 1
Not completed — Parents personal problem | 0 | 0 | 1
Not completed — Subject eliminated (other vaccine) | 1 | 0 | 0
Not completed — Withdrawal by Subject | 3 | 0 | 2
Not completed — Lost to Follow-up | 8 | 8 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Priorix-Tetra Group | Priorix/ Priorix-Tetra Group | Control Group | Total
Number analyzed (Participants) | 180 | 180 | 90 | 450
Age, Continuous [Mean (Standard Deviation); unit: Months] | 9 (0) | 9 (0.11) | 9 (0) | 9 (0.07)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 79 | 89 | 49 | 217
  Male | 101 | 91 | 41 | 233
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian - central/ south Asian heritage | 177 | 175 | 88 | 440
  Asian - south east Asian heritage | 2 | 5 | 2 | 9
  American Indian or Alaskan native | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Seroconverted for Measles, Mumps, Rubella and Varicella Antibodies
Description: Seroconversion was defined as the appearance of antibodies [i.e. concentration/titre greater than or equal to (≥) the cut-off value] in the serum of subjects seronegative before vaccination. The cut-off values for seroconversion were 150 milli-international units per milliliter (mIU/mL), 231 units per milliliter (U/mL), 4 international units per milliliter (IU/mL) and for immunoglobulin G (IgG) varicella antibodies 1:4 dilution for measles, mumps, rubella and varicella, respectively.
Time Frame: At 42 - 56 days after the second vaccination dose at week 30
Population: The analysis was performed on the According-To-Protocol (ATP) cohort for immunogenicity, which included all eligible subjects for whom pre-vaccination and post-vaccination serology results were available for antibodies against at least one antigen.
Measure: Count of Participants; unit: Participants
Arm/Group | Priorix-Tetra Group | Priorix/ Priorix-Tetra Group | Control Group
Number analyzed (Participants) | 150 | 153 | 73
Participants
  Anti-measles ≥ 150 mIU/mL: number analyzed (Participants) | 149 | 153 | 72
  Anti-measles ≥ 150 mIU/mL | 149 | 153 | 72
  Anti-mumps ≥ 231 U/ML: number analyzed (Participants) | 149 | 152 | 72
  Anti-mumps ≥ 231 U/ML | 149 | 152 | 72
  Anti-rubella ≥ 4 IU/mL: number analyzed (Participants) | 150 | 152 | 73
  Anti-rubella ≥ 4 IU/mL | 150 | 152 | 73
  IgG varicella antibodies ≥ 1:4: number analyzed (Participants) | 138 | 143 | 72
  IgG varicella antibodies ≥ 1:4 | 138 | 141 | 69
Statistical Analysis 1: Comparison: Priorix-Tetra Group vs Control Group; Non-inferiority of 2 doses of Priorix-Tetra® vaccine compared to Priorix™ vaccine followed by Priorix™ vaccine co-administered with Varilrix™ vaccine in terms of anti-measles seroconversion rates; Test type: Non-Inferiority — Non-inferiority with respect to seroconversion rates for measles 42-56 days after second vaccination dose was concluded if the lower limit (LL) of the two-sided standardised asymptotic 95% CI on the difference in the seroconversion rates between the two groups (Priorix-Tetra Group minus Control Group) was greater than or equal to (≥) -10%; Difference in percentage = 0, 95% CI 2-sided [-2.52 to 5.09]
Statistical Analysis 2: Comparison: Priorix-Tetra Group vs Control Group; Non-inferiority of 2 doses of Priorix-Tetra® vaccine compared to Priorix™ vaccine followed by Priorix™ vaccine co-administered with Varilrix™ vaccine in terms of anti-mumps seroconversion rates; Test type: Non-Inferiority — Non-inferiority with respect to seroconversion rates for mumps 42-56 days after second vaccination dose was concluded if the lower limit (LL) of the two-sided standardised asymptotic 95% CI on the difference in the seroconversion rates between the two groups (Priorix-Tetra Group minus Control Group) was greater than or equal to (≥) -10%; Difference in percentage = 0, 95% CI 2-sided [-2.52 to 5.09]
Statistical Analysis 3: Comparison: Priorix-Tetra Group vs Control Group; Non-inferiority of 2 doses of Priorix-Tetra® vaccine compared to Priorix™ vaccine followed by Priorix™ vaccine co-administered with Varilrix™ vaccine in terms of anti-rubella seroconversion rates; Test type: Non-Inferiority — Non-inferiority with respect to seroconversion rates for rubella 42-56 days after second vaccination dose was concluded if the lower limit (LL) of the two-sided standardised asymptotic 95% CI on the difference in the seroconversion rates between the two groups (Priorix-Tetra Group minus Control Group) was greater than or equal to (≥) -10%; Difference in percentage = 0, 95% CI 2-sided [-2.51 to 5.02]
Statistical Analysis 4: Comparison: Priorix-Tetra Group vs Control Group; Non-inferiority of 2 doses of Priorix-Tetra® vaccine compared to Priorix™ vaccine followed by Priorix™ vaccine co-administered with Varilrix™ vaccine in terms of anti-varicella seroconversion rates; Test type: Non-Inferiority — Non-inferiority with respect to seroconversion rates for varicella 42-56 days after second vaccination dose was concluded if the lower limit (LL) of the two-sided standardised asymptotic 95% CI on the difference in the seroconversion rates between the two groups (Priorix-Tetra Group minus Control Group) was greater than or equal to (≥) -10%; Difference in percentage = 4.17, 95% CI 2-sided [1.37 to 11.57]
Statistical Analysis 5: Comparison: Priorix/ Priorix-Tetra Group vs Control Group; Non-inferiority of Priorix™ vaccine followed by Priorix-Tetra® vaccine compared to Priorix™ vaccine followed by Priorix™ vaccine co-administered with Varilrix™ vaccine in terms of anti-measles seroconversion rates; Test type: Non-Inferiority — Non-inferiority with respect to seroconversion rates for measles 42-56 days after second vaccination dose was concluded if the lower limit (LL) of the 2-sided standardised asymptotic 95% confidence interval (CI) on the difference in the seroconversion rates between the 2 groups (Priorix/Priorix-Tetra Group minus Control Group) was ≥ -10%; Difference in percentage = 0, 95% CI 2-sided [-2.46 to 5.09]
Statistical Analysis 6: Comparison: Priorix/ Priorix-Tetra Group vs Control Group; Non-inferiority of Priorix™ vaccine followed by Priorix-Tetra® vaccine compared to Priorix™ vaccine followed by Priorix™ vaccine co-administered with Varilrix™ vaccine in terms of anti-mumps seroconversion rates; Test type: Non-Inferiority — Non-inferiority with respect to seroconversion rates for mumps 42-56 days after second vaccination dose was concluded if the lower limit (LL) of the 2-sided standardised asymptotic 95% confidence interval (CI) on the difference in the seroconversion rates between the 2 groups (Priorix/Priorix-Tetra Group minus Control Group) was ≥ -10%; Difference in percentage = 0, 95% CI 2-sided [-2.48 to 5.09]
Statistical Analysis 7: Comparison: Priorix/ Priorix-Tetra Group vs Control Group; Non-inferiority of Priorix™ vaccine followed by Priorix-Tetra® vaccine compared to Priorix™ vaccine followed by Priorix™ vaccine co-administered with Varilrix™ vaccine in terms of anti-rubella seroconversion rates; Test type: Non-Inferiority — Non-inferiority with respect to seroconversion rates for rubella 42-56 days after second vaccination dose was concluded if the lower limit (LL) of the 2-sided standardised asymptotic 95% confidence interval (CI) on the difference in the seroconversion rates between the 2 groups (Priorix/Priorix-Tetra Group minus Control Group) was ≥ -10%; Difference in percentage = 0, 95% CI 2-sided [-2.48 to 5.02]
Statistical Analysis 8: Comparison: Priorix/ Priorix-Tetra Group vs Control Group; Non-inferiority of Priorix™ vaccine followed by Priorix-Tetra® vaccine compared to Priorix™ vaccine followed by Priorix™ vaccine co-administered with Varilrix™ vaccine in terms of anti-varicella seroconversion rates; Test type: Non-Inferiority — Non-inferiority with respect to seroconversion rates for varicella 42-56 days after second vaccination dose was concluded if the lower limit (LL) of the 2-sided standardised asymptotic 95% confidence interval (CI) on the difference in the seroconversion rates between the 2 groups (Priorix/Priorix-Tetra Group minus Control Group) was ≥ -10%; Difference in percentage = 2.77, 95% CI 2-sided [-1.59 to 10.29]

2. Secondary Outcome: Number of Seroconverted Subjects for Measles, Mumps, Rubella and Varicella Antibodies
Description: Seroconversion was defined as the appearance of antibodies (i.e. concentration/titre ≥ the cut-off value) in the serum of subjects seronegative before vaccination. The cut-off values for seroconversion were 150 mIU/mL, 231 U/mL, 4 IU/mL and for IgG varicella antibodies 1:4 dilution for measles, mumps, rubella and varicella, respectively.
Time Frame: Approximately 42 to 56 days after the first vaccine dose at week 6
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Priorix-Tetra Group | Priorix/ Priorix-Tetra Group | Control Group
Number analyzed (Participants) | 149 | 153 | 73
Participants
  Anti-measles ≥ 150 mIU/mL: number analyzed (Participants) | 148 | 153 | 72
  Anti-measles ≥ 150 mIU/mL | 138 | 135 | 63
  Anti-mumps ≥ 231 U/ML: number analyzed (Participants) | 144 | 152 | 72
  Anti-mumps ≥ 231 U/ML | 124 | 128 | 60
  Anti-rubella ≥ 4 IU/mL: number analyzed (Participants) | 149 | 152 | 73
  Anti-rubella ≥ 4 IU/mL | 147 | 151 | 73
  IgG varicella antibodies ≥ 1:4: number analyzed (Participants) | 138 | 142 | 72
  IgG varicella antibodies ≥ 1:4 | 130 | 4 | 1

3. Secondary Outcome: Antibody Concentrations Against Measles, Mumps, Rubella and Varicella Viruses
Description: Antibody concentrations were summarized by geometric mean concentrations (GMCs) with their 95% confidence intervals (CIs).
Time Frame: At 42 - 56 days after the first (at Week 6) and second (at Week 30) vaccination dose
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | Priorix-Tetra Group | Priorix/ Priorix-Tetra Group | Control Group
Number analyzed (Participants) | 150 | 153 | 73
mIU/mL
  Anti-measles; Week 6: number analyzed (Participants) | 148 | 153 | 72
  Anti-measles; Week 6 | 2013.6 [1662.2 to 2439.3] | 1180.4 [963 to 1446.7] | 1200 [887.9 to 1621.8]
  Anti-mumps; Week 6: number analyzed (Participants) | 144 | 152 | 72
  Anti-mumps; Week 6 | 991.9 [819.7 to 1200.3] | 746.6 [628 to 887.6] | 775.1 [600.9 to 999.7]
  Anti-rubella; Week 6: number analyzed (Participants) | 149 | 152 | 73
  Anti-rubella; Week 6 | 45.4 [38.3 to 53.7] | 63.8 [55.9 to 72.8] | 62 [51.3 to 74.9]
  IgG varicella antibodies; Week 6: number analyzed (Participants) | 138 | 142 | 72
  IgG varicella antibodies; Week 6 | 120.5 [90.8 to 160] | 2.2 [2 to 2.4] | 2.2 [1.8 to 2.6]
  Anti-measles; Week 30: number analyzed (Participants) | 149 | 153 | 72
  Anti-measles; Week 30 | 4471.3 [3975.3 to 5029.2] | 3358.7 [3017.5 to 3738.4] | 2495 [2064.5 to 3015.2]
  Anti-mumps; Week 30: number analyzed (Participants) | 149 | 152 | 72
  Anti-mumps; Week 30 | 6428 [5774.9 to 7154.9] | 10108.5 [9223.9 to 11078] | 4925.3 [4200.9 to 5774.7]
  Anti-rubella; Week 30: number analyzed (Participants) | 150 | 152 | 73
  Anti-rubella; Week 30 | 148.4 [136.1 to 161.8] | 164.8 [152.1 to 178.6] | 173 [153 to 195.6]
  IgG varicella antibodies; Week 30: number analyzed (Participants) | 138 | 143 | 72
  IgG varicella antibodies; Week 30 | 5318.5 [4318.7 to 6549.8] | 198 [158.2 to 247.7] | 128 [91.7 to 178.7]

4. Secondary Outcome: Number of Subjects Reporting Any and Grade 3 Solicited Local Symptoms
Description: Assessed solicited local symptoms were pain, redness and swelling. Any = occurrence of the symptom regardless of intensity grade. Grade 3 pain = cried when limb was moved/spontaneously painful. Grade 3 redness/swelling = redness/swelling spreading beyond 20 millimeters (mm) of injection site.
Time Frame: During the 4-day (Days 0-3) post-vaccination period following each dose (Dose 1 and Dose 2)
Population: The analysis was performed on the Total Vaccinated cohort, which included all vaccinated subjects with the symptom sheet filled in.
Measure: Count of Participants; unit: Participants
Arm/Group | Priorix-Tetra Group | Priorix/ Priorix-Tetra Group | Control Group
Number analyzed (Participants) | 174 | 172 | 84
Participants
  Any Pain; Dose 1 | 20 | 12 | 9
  Grade 3 Pain; Dose 1 | 0 | 0 | 0
  Any Redness; Dose 1 | 15 | 8 | 3
  Grade 3 Redness; Dose 1 | 0 | 0 | 0
  Any Swelling; Dose 1 | 8 | 5 | 3
  Grade 3 Swelling; Dose 1 | 0 | 0 | 0
  Any Pain; Dose 2: number analyzed (Participants) | 155 | 159 | 79
  Any Pain; Dose 2 | 9 | 10 | 3
  Grade 3 Pain; Dose 2: number analyzed (Participants) | 155 | 159 | 79
  Grade 3 Pain; Dose 2 | 0 | 0 | 0
  Any Redness; Dose 2: number analyzed (Participants) | 155 | 159 | 79
  Any Redness; Dose 2 | 10 | 6 | 0
  Grade 3 Redness; Dose 2: number analyzed (Participants) | 155 | 159 | 79
  Grade 3 Redness; Dose 2 | 3 | 0 | 0
  Any Swelling; Dose 2: number analyzed (Participants) | 155 | 159 | 79
  Any Swelling; Dose 2 | 9 | 6 | 0
  Grade 3 Swelling; Dose 2: number analyzed (Participants) | 155 | 159 | 79
  Grade 3 Swelling; Dose 2 | 0 | 0 | 0

5. Secondary Outcome: Number of Subjects Reporting Any, Grade 3 and Related Solicited General Symptoms
Description: Assessed solicited general symptoms were meningism and parotid gland swelling. Any = occurrence of the symptom regardless of intensity grade or relationship to vaccination. Grade 3 meningism and parotid gland swelling = meningism/parotid gland swelling which prevented normal everyday activities. Related = symptom assessed by the investigator as related to the vaccination.
Time Frame: During the 43-day (Days 0-42) post-vaccination period following each dose (Dose 1 and Dose 2)
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Priorix-Tetra Group | Priorix/ Priorix-Tetra Group | Control Group
Number analyzed (Participants) | 174 | 172 | 83
Participants
  Any Meningism; Dose 1 | 0 | 0 | 0
  Grade 3 Meningism; Dose 1 | 0 | 0 | 0
  Related Meningism; Dose 1 | 0 | 0 | 0
  Any Parotid gland swelling; Dose 1 | 0 | 0 | 0
  Grade 3 Parotid gland swelling; Dose 1 | 0 | 0 | 0
  Related Parotid gland swelling; Dose 1 | 0 | 0 | 0
  Any Meningism; Dose 2: number analyzed (Participants) | 155 | 159 | 79
  Any Meningism; Dose 2 | 0 | 0 | 0
  Grade 3 Meningism; Dose 2: number analyzed (Participants) | 155 | 159 | 79
  Grade 3 Meningism; Dose 2 | 0 | 0 | 0
  Related Meningism; Dose 2: number analyzed (Participants) | 155 | 159 | 79
  Related Meningism; Dose 2 | 0 | 0 | 0
  Any Parotid gland swelling; Dose 2: number analyzed (Participants) | 155 | 159 | 79
  Any Parotid gland swelling; Dose 2 | 0 | 0 | 0
  Grade 3 Parotid gland swelling; Dose 2: number analyzed (Participants) | 155 | 159 | 79
  Grade 3 Parotid gland swelling; Dose 2 | 0 | 0 | 0
  Related Parotid gland swelling; Dose 2: number analyzed (Participants) | 155 | 159 | 79
  Related Parotid gland swelling; Dose 2 | 0 | 0 | 0

6. Secondary Outcome: Number of Subjects Reporting Any, Grade 3 and Related Fever
Description: Any fever was defined as fever ≥ 38.0°C and grade 3 fever was defined as fever > 39.5°C after vaccination. Related fever was defined as fever assessed by the investigator as related to the vaccination.
Time Frame: During the 43-day (Days 0-42) post-vaccination period following each dose (Dose 1 and Dose 2)
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Priorix-Tetra Group | Priorix/ Priorix-Tetra Group | Control Group
Number analyzed (Participants) | 174 | 172 | 83
Participants
  Any temperature; Dose 1 | 76 | 70 | 27
  Grade 3 temperature; Dose 1 | 11 | 5 | 1
  Related temperature; Dose 1 | 53 | 48 | 15
  Any temperature; Dose 2: number analyzed (Participants) | 155 | 159 | 79
  Any temperature; Dose 2 | 41 | 37 | 22
  Grade 3 temperature; Dose 2: number analyzed (Participants) | 155 | 159 | 79
  Grade 3 temperature; Dose 2 | 2 | 6 | 2
  Related temperature; Dose 2: number analyzed (Participants) | 155 | 159 | 79
  Related temperature; Dose 2 | 22 | 21 | 10

7. Secondary Outcome: Number of Subjects Reporting Any, Grade 3 and Related Rash
Description: Any rash was defined as incidence of a rash regardless of intensity grade or relationship to vaccination and grade 3 rash greater than (>) 150 lesions. Related rash was defined as rash assessed by the investigator as causally related to the vaccination
Time Frame: During the 43-day (Days 0-42) post-vaccination period following each dose (Dose 1 and Dose 2)
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Priorix-Tetra Group | Priorix/ Priorix-Tetra Group | Control Group
Number analyzed (Participants) | 174 | 172 | 83
Participants
  Any Rash; Dose 1 | 1 | 2 | 1
  Grade 3 Rash; Dose 1 | 0 | 0 | 0
  Related Rash; Dose 1 | 1 | 0 | 0
  Any Rash; Dose 2: number analyzed (Participants) | 155 | 159 | 79
  Any Rash; Dose 2 | 0 | 1 | 0
  Grade 3 Rash; Dose 2: number analyzed (Participants) | 155 | 159 | 79
  Grade 3 Rash; Dose 2 | 0 | 0 | 0
  Related Rash; Dose 2: number analyzed (Participants) | 155 | 159 | 79
  Related Rash; Dose 2 | 0 | 0 | 0

8. Secondary Outcome: Number of Subjects Reporting Any Unsolicited Adverse Event
Description: An unsolicited Adverse Event (AE) covers any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. Any was defined as an AE reported in addition to those solicited during the clinical study. Also any 'solicited' symptom with onset outside the specified period of follow-up for solicited symptoms was reported as an unsolicited adverse event.
Time Frame: Within 43-day (Days 0-42) after the first and second vaccination dose
Population: The analysis was performed on the Total Vaccinated cohort, which included all vaccinated subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | Priorix-Tetra Group | Priorix/ Priorix-Tetra Group | Control Group
Number analyzed (Participants) | 180 | 180 | 90
Participants
  Any AE(s); Dose 1 | 37 | 39 | 18
  Any AE(s); Dose 2 | 19 | 18 | 11

9. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs)
Description: Serious adverse events (SAEs) assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization, result in disability/incapacity or congenital anomaly/birth defect in the offspring of a study subject.
Time Frame: From the first study dose up to study end (Month 0 to Month 7.5 approximately)
Population: The analysis was performed on the Total Vaccinated cohort, which included all vaccinated subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | Priorix-Tetra Group | Priorix/ Priorix-Tetra Group | Control Group
Number analyzed (Participants) | 180 | 180 | 90
Participants | 7 | 6 | 0

ADVERSE EVENTS:
Time Frame: Solicited local and general symptoms were collected during the 4-day and 43-day after each vaccination dose respectively. Unsolicited AEs were collected during the 43-day after each vaccination dose. SAEs were collected from Month 0 to Month 7.5.
Arm/Group | Priorix-Tetra Group | Priorix/ Priorix-Tetra Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/180 | 0/180 | 0/90
Serious Adverse Events (participants affected / at risk) | 7/180 | 6/180 | 0/90
Other Adverse Events (participants affected / at risk) | 114/180 | 116/180 | 55/90
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Priorix-Tetra Group (N=180) | Priorix/ Priorix-Tetra Group (N=180) | Control Group (N=90)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Febrile convulsion (Nervous system disorders) | 0 | 1 | 0
Pyrexia (General disorders) | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 2 | 3 | 0
Lower respiratory tract infection (Infections and infestations) | 2 | 1 | 0
Viral infection (Infections and infestations) | 1 | 1 | 0
Bronchiolitis (Infections and infestations) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Priorix-Tetra Group (N=180) | Priorix/ Priorix-Tetra Group (N=180) | Control Group (N=90)
Cough; Dose 1 (Respiratory, thoracic and mediastinal disorders) | 6 | 10 | 6
Pain; Dose 1 (General disorders) | 20 | 12 | 9
Redness; Dose 1 (General disorders) | 15/174 | 8/172 | 3/84
Pain; Dose 2 (General disorders) | 9/155 | 10/159 | 3/79
Redness; Dose 2 (General disorders) | 10/155 | 6/159 | 0/79
Swelling; Dose 2 (General disorders) | 9/155 | 6/159 | 0/79
Fever; Dose 1 (General disorders) | 76/174 | 70/172 | 27/83
Fever; Dose 2 (General disorders) | 41/155 | 37/159 | 22/79
Rhinitis; Dose 1 (Infections and infestations) | 7 | 9 | 6
Nasopharyngitis; Dose 1 (Infections and infestations) | 4 | 8 | 6
Upper respiratory tract infection; Dose 1 (Infections and infestations) | 10 | 7 | 1
Rhinitis; Dose 2 (Infections and infestations) | 6 | 7 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.